CLINICAL TRIAL: NCT02533206
Title: Endoscopic Polypectomy Performed In Clinic (EPIC) for Chronic Rhinosinusitis With Polyps: Pilot Study of The EPIC Randomised Controlled Trial
Brief Title: Pilot Study of The EPIC Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150487-01H
Record Dates: First submitted 2015-07-06; First posted 2015-08-26 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Sinusitis; Nasal Polyps
MeSH Terms: conditions — Sinusitis; Nasal Polyps | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPIC (Experimental): The experimental intervention is endoscopic polypectomy performed in clinic (EPIC) where nasal polyps are removed using a microdebrider under local and topical anesthesia in the outpatient clinic. The participant will be discharged home from the clinic following their procedure.
  Interventions: Procedure: Endoscopic Polypectomy Performed in Clinic
- FESS (Active Comparator): The control intervention is functional endoscopic sinus surgery (FESS), a minimally invasive procedure that is the current standard that involves polypectomy with a microdebrider as well as sinus ostia enlargement of the affected sinuses performed in the operating room under general anesthesia
  Interventions: Procedure: Functional Endoscopic Sinus Surgery (FESS)

INTERVENTIONS:
Procedure: Endoscopic Polypectomy Performed in Clinic — Endoscopic polypectomy performed in clinic under local and topical anesthesia
  Other Names: EPIC
  Arms: EPIC
Procedure: Functional Endoscopic Sinus Surgery (FESS) — Functional Endoscopic Sinus Surgery
  Other Names: FESS
  Arms: FESS

SUMMARY:
Chronic sinusitis is one of the most common chronic diseases in North America, with over 5% of the Canadian population affected by the disease. Until now, treatment with surgery has been performed only in the operating room. Recently a smaller surgical procedure that is done in the clinic for some patients with chronic sinusitis with polyps has been found to result in symptom control that appears to be similar to that which occurs with sinus surgery. Performing the smaller clinical procedure has advantages including a shorter recovery time for the patient, a much lower cost to the health care system for the procedure, and a shorter patient wait time for the procedure to be done in comparison to sinus surgery performed in the operating room. To know with greater certainty that the procedure performed in the clinic is as good as the operating room sinus surgery, a large multiple investigator randomised clinical trial has been designed. However, before carrying out that trial, a practice run or internal pilot study of that trial is required to ensure that the trial can recruit patients at the rate that is anticipated and that the procedures to obtain the measurements being used for the larger study are adequate.

DETAILED DESCRIPTION:
For the proposed internal pilot study 20 patients who consent to participate and meet all inclusion criteria and none of the inclusion criteria will be enrolled. The internal pilot study will be carried out at sites located in Ottawa , Winchester, Toronto, Barrie, Sault Saint Marie and London Ontario. A total of 7 investigator-surgeons will participate. Since this is an internal pilot study a sample size was not calculated, rather, the 20 patients enrolled in the internal pilot study will be included as part of the total sample of the definite non-inferiority trial, which has been calculated to be 140 patients. The pilot will recruit 15% of the total sample which is sufficient to achieve the main goal of this pilot i.e. establish the feasibility of the main trial. Eligible participants will be randomly assigned in a 1:1 fashion to either the experimental (endoscopic polypectomy performed in clinic, EPIC) or the control group (functional endoscopic sinus surgery, FESS) . Patients will be allocated to treatment group using web-based central randomization to protect against bias , these data will be used to confirm the design the non-inferiority randomized control trial.

Duration of treatment period For both experimental (endoscopic polypectomy performed in clinic, EPIC) and control (functional endoscopic sinus surgery, FESS) groups, the day the treatment is completed will be considered to be time "0". There is no change to either procedure related to the participant having enrolled into the study. After the treatment day, participants will enter a follow-up period where the final study related evaluation is 90(± 5) days following their procedure.

Frequency and duration of follow up Enrolled participants will be re-evaluated by the investigators after their procedure twice, which is the normal frequency of visits for postoperative care for patients who have undergone surgical treatment for chronic rhinosinusitis with polyps. The first follow-up evaluation at 15 days (± 5 days) following the procedure and the last will occur 90 days (± 5 days) following the treatment. The last follow-up is chosen to be at 90 days given the primary outcome measure of interest is the sinonasal outcome test-22 (SNOT-22) score. Three months after treatment the SNOT-22 does not appear to change substantially with further follow-up. A landmark study completed by Hopkins et al. (2006) with a cohort of over 3000 patients who had undergone endoscopic sinus surgery for chronic sinusitis and who were followed for 36 months demonstrated that the sinonasal outcome test SNOT-22 scores at 3 months following surgery were not different from those measured at 12 or 36 months. Therefore, the 3-month (90 days) follow-up has been specifically chosen for this study given the primary outcome measure being used is also the SNOT-22 score.

Long Term Follow up:

After the second follow up visit, patients will enter a long term follow-up period which will last 5 years. During this period, patients will receive the following questionnaires via mail: SNOT-22, EuroQol (EQ-5D-5L) questionnaire, work productivity and impairment questionnaire (WPAI), Satisfaction Survey and the Individual Health Resource Consumption. These questionnaires will be mailed at 6 months, 1,2,3,4 and 5 years after the procedure. At this time patients will also be asked if they have had additional surgeries for their chronic rhinosinusitis with nasal polyps

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Diagnosis of chronic rhinosinusitis with polyps requiring surgical treatment after having been treated with medical therapy as designated by the Canadian clinical practice guidelines for acute and chronic sinusitis. 21
3. Bilateral nasal polyps present of Grade ≥ 2 on each side as determined by the Lildholdt scale score measured by nasal endoscopy (Appendix 2) at the screening visit.
4. Must have nasal blockage score greater than or equal to 4 on the sinonasal outcome test SNOT-22 (Appendix 3) at the screening visit.
5. Must have an American Society of Anesthesiologists physical status (ASA PS) 3 classification or less. ASA PS 3: Patients with severe systemic disease: Some functional limitation; has a controlled disease of more than one body system or one major system; no immediate danger of death. ASA PS 2: Patients with mild systemic disease. No functional limitations; has a well-controlled disease of one body system. ASA PS 1: Normal healthy patient. No organic, physiologic, or psychiatric disturbance; excludes the very young and very old.
6. Participants with comorbid asthma or chronic obstructive pulmonary disease (COPD) must have stable disease with no exacerbations (no emergency room visits, hospitalisations, or oral or parental steroid use for these lower respiratory conditions) within 3 months before the screening visit.
7. Must be capable, in the opinion of the investigator, of providing informed consent to participate in the study. Participants must sign an informed consent document indicating that they understand the purpose of and procedures of the study and are willing to participate in the study.

Exclusion Criteria:

1. Women who are pregnant or breast feeding
2. Patients with hyperplastic polyps or polyps large enough that they result in external nasal deformity
3. Facial pain/pressure score higher than 2 on the sinonasal outcome test SNOT-22 at the screening visit.
4. History of any surgical procedure that prevents the ability to accurately grade the nasal polyps
5. Participants who will not be able to complete the follow-up appointments/evaluations
6. Have significant oral structural abnormalities, e.g. unrepaired cleft palate
7. Septal deviation requiring correction in order to perform either EPIC or FESS procedures
8. Diagnosis of an immunodeficiency or immunocompromised state
9. Diagnosis of cystic fibrosis
10. Diagnosis of allergic fungal sinusitis
11. Contraindication to the use of oral corticosteroids (e.g. uncontrolled diabetes, congestive heart failure, uncontrolled hypertension, known renal insufficiency, known peptic ulcer disease, known glaucoma, pregnancy)
12. History of either Churg-Strauss syndrome, primary ciliary dyskinesia, or vasculitis (e.g. granulomatosis with polyangiitis(GPA))
13. Allergy, hypersensitivity, or contraindication to the use of local or topical lidocaine anesthetics, nasal topical 1:1000 adrenaline, nasal decongestants, nasal steroid spray
14. Any serious or unstable concurrent disease, psychiatric disorder, or any significant condition that, in the opinion of the investigator, could confound the results of the study or could interfere with the participant's participation or compliance with the study
15. A recent (within 1 year of the screening visit) clinically significant history of drug or alcohol abuse, or dependence that, in the opinion of the investigator could interfere with the participant's participation or compliance with the study
16. Inability to read and understand English
17. Any medical condition that in the opinion of the investigator would interfere with the treatment
18. Any participant who is unfit to undergo surgery under general anesthesia
19. Current participation in another clinical trial at the time of the screening visit.
20. Participant is unable to undergo an awake procedure
21. Diagnosis or Aspirin Exacerbated Respiratory Disease (AERD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-08; Primary Completion 2022-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment | One year
  Number of patients recruited in one year

SECONDARY OUTCOMES:
Arm cross-over | One year
  Number of participants who switched arm
Loss to follow up | Evaluated at 6 months after intervention
  Number of participants who do not complete the 6 month follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Kilty, MD, FRCSC, Principal Investigator — The Ottawa Hospital Research Institute
Locations (5):
- Canada (5):
  - Royal Victoria Hospital, Barrie, Ontario
  - St Joseph's Health Care, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Algoma District Medical Group, Sault Ste. Marie, Ontario
  - Saint Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Background] Rudmik L, Smith KA, Kilty S. Endoscopic polypectomy in the clinic: a pilot cost-effectiveness analysis. Clin Otolaryngol. 2016 Apr;41(2):110-7. doi: 10.1111/coa.12473. Epub 2016 Feb 4. PMID 26053107
- [Background] Kilty SJ. In-clinic endoscopic polypectomy for chronic rhinosinusitis with polyps: a treatment strategy pilot study in ten adults. Clin Otolaryngol. 2015 Jun;40(3):281-4. doi: 10.1111/coa.12372. No abstract available. PMID 25581621